CLINICAL TRIAL: NCT00754130
Title: A Multiple Dose Study to Assess the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of MK-0941 in Japanese Patients With Type 2 Diabetes
Brief Title: MK-0941 Multiple Dose Study in Japanese Patients With Type 2 Diabetes (MK-0941-011).
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0941-011; 2008_023 (Other: Merck Registration ID); MK-0941-011 (Other: Merck Protocol ID)
Record Dates: First submitted 2008-09-16; First posted 2008-09-17 (Estimated); Results first posted 2012-10-03 (Estimated); Last update posted 2015-03-12 (Estimated); Status verified 2015-02

CONDITIONS: Diabetes Mellitus, Non-Insulin-Dependent
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — 3-((6-(ethylsulfonyl)-3-pyridinyl)oxy)-5-(2-hydroxy-1-methylethoxy)-N-(1-methyl-1H-pyrazol-3-yl)benzamide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (6):
- Placebo/MK-0941 20mg (Experimental): Participants received Placebo during Period 1 and MK-0941 20 mg during Period 2. There was a washout period of at least 8 days between the two treatment periods.
  Interventions: Drug: Placebo; Drug: MK-0941
- MK-0941 5mg/Placebo (Experimental): Participants received MK-0941 5 mg during Period 1 and Placebo during Period 2. There was a washout period of at least 8 days between the two treatment periods.
  Interventions: Drug: Placebo; Drug: MK-0941
- MK-0941 5mg/MK-0941 20mg (Experimental): Participants received MK-0941 5 mg during Period 1 and MK-0941 20 mg during Period 2. There was a washout period of at least 8 days between the two treatment periods.
  Interventions: Drug: MK-0941
- Placebo/MK-0941 40mg (Experimental): Participants received Placebo during Period 1 and MK-0941 40 mg during Period 2. There was a washout period of at least 8 days between the two treatment periods.
  Interventions: Drug: Placebo; Drug: MK-0941
- MK-0941 10mg/Placebo (Experimental): Participants received MK-0941 10 mg during Period 1 and Placebo during Period 2. There was a washout period of at least 8 days between the two treatment periods.
  Interventions: Drug: Placebo; Drug: MK-0941
- MK-0941 10mg/MK-0941 40mg (Experimental): Participants received MK-0941 10 mg during Period 1 and MK-0941 40 mg during Period 2. There was a washout period of at least 8 days between the two treatment periods.
  Interventions: Drug: MK-0941

INTERVENTIONS:
Drug: Placebo — Placebo tablets before every meal (q.a.c) Treatment period is 5 days.
  Arms: MK-0941 10mg/Placebo; MK-0941 5mg/Placebo; Placebo/MK-0941 20mg; Placebo/MK-0941 40mg
Drug: MK-0941 — MK-0941 5 mg tablets q.a.c.; 10 mg tablets q.a.c.; 20 mg tablets q.a.c.; or 40 mg tablets q.a.c. Treatment period is 5 days.

SUMMARY:
The multiple dose study to assess the safety, tolerability, pharmacokinetics and pharmacodynamics of MK-0941 in Japanese patients with Type 2 Diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Japanese Male or Female between 20 to 65 years of age
* Diagnosis of Type 2 Diabetes
* Patient being treated by diet and exercise alone

Exclusion Criteria:

* Patient has a history of Type 1 Diabetes
* Patient is being treated with glaucoma medications
* Patient has donated blood or participated in another clinical study in the past 12 weeks
* Patient is a regular user of any illicit drugs or has a history of drug, including alcohol, abuse

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2008-09; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo/MK-0941 20mg: Participants received Placebo during Period 1 and MK-0941 20 mg during Period 2
- MK-0941 5mg/Placebo: Participants received MK-0941 5 mg during Period 1 and Placebo during Period 2
- MK-0941 5mg/MK-0941 20mg: Participants received MK-0941 5 mg during Period 1 and MK-0941 20 mg during Period 2
- Placebo/MK-0941 40mg: Participants received Placebo during Period 1 and MK-0941 40 mg during Period 2
- MK-0941 10mg/Placebo: Participants received MK-0941 10 mg during Period 1 and Placebo during Period 2
- MK-0941 10mg/MK-0941 40mg: Participants received MK-0941 10 mg during Period 1 and MK-0941 40 mg during Period 2
Period: Period 1 (5 Days)
Arm/Group | Placebo/MK-0941 20mg | MK-0941 5mg/Placebo | MK-0941 5mg/MK-0941 20mg | Placebo/MK-0941 40mg | MK-0941 10mg/Placebo | MK-0941 10mg/MK-0941 40mg
Started | 2 | 2 | 4 | 2 | 2 | 4 (One participant received MK-0941 10 mg in both Periods 1 and 2.)
Completed | 2 | 2 | 4 | 2 | 2 | 4
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Washout Period (>=8 Days)
Arm/Group | Placebo/MK-0941 20mg | MK-0941 5mg/Placebo | MK-0941 5mg/MK-0941 20mg | Placebo/MK-0941 40mg | MK-0941 10mg/Placebo | MK-0941 10mg/MK-0941 40mg
Started | 2 | 2 | 4 | 2 | 2 | 4
Completed | 2 | 2 | 4 | 2 | 2 | 4
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Period 2 (5 Days)
Arm/Group | Placebo/MK-0941 20mg | MK-0941 5mg/Placebo | MK-0941 5mg/MK-0941 20mg | Placebo/MK-0941 40mg | MK-0941 10mg/Placebo | MK-0941 10mg/MK-0941 40mg
Started | 2 (One participant received MK-0941 15 mg starting with Dose 2 on Day 2.) | 2 | 4 | 2 | 2 | 4 (One participant received MK-0941 35 mg starting with Dose 3 on Day 3.)
Completed | 2 | 2 | 4 | 2 | 2 | 4
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo/MK-0941 20mg | MK-0941 5mg/Placebo | MK-0941 5mg/MK-0941 20mg | Placebo/MK-0941 40mg | MK-0941 10mg/Placebo | MK-0941 10mg/MK-0941 40mg | Total
Number analyzed (Participants) | 2 | 2 | 4 | 2 | 2 | 4 | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.0 (12.73) | 48.5 (2.12) | 45.5 (16.58) | 57.0 (7.07) | 53.5 (10.60) | 51.5 (11.36) | 50.4 (10.82)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 1 | 0 | 1 | 2
  Male | 2 | 2 | 4 | 1 | 2 | 3 | 14

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Experienced at Least One Adverse Event (AE)
Description: An AE is defined as any unfavorable and unintended change in the structure, function, or chemistry of the body temporally associated with the use of the study drug, whether or not considered related to the use of the product.
  Participants were monitored for occurrence AEs for up to 8 days after last dose of study drug during Period 1 and for up to 14 days after last dose of study drug during Period 2.
Time Frame: Up to 14 days after last dose of study drug
Population: Safety Population, consisting of all randomized participants who received at least one dose of study drug.
Measure: Number; unit: participants
Groups:
- Placebo: Participants receiving Placebo doses three times daily
- MK-0941 5mg: Participants receiving MK-0941 5 mg doses three times daily
- MK-0941 10mg: Participants receiving MK-0941 10 mg doses three times daily
- MK-0941 20mg: Participants receiving MK-0941 20 mg doses three times daily
- MK-0941 40mg: Participants receiving MK-0941 40 mg doses three times daily. One participant randomized to receive MK-0941 10 mg during Period 1 and MK-0941 40 mg during Period 2 received MK-0941 10 mg during both Periods 1 and 2.
Arm/Group | Placebo | MK-0941 5mg | MK-0941 10mg | MK-0941 20mg | MK-0941 40mg
Number analyzed (Participants) | 8 | 6 | 6 | 6 | 5
participants | 2 | 2 | 2 | 2 | 2

2. Secondary Outcome: Plasma Pharmacokinetic Parameter: Area Under the Concentration-time Curve (AUC)(0-24hr) of MK-0941
Description: Blood samples for measurement of plasma pharmacokinetic parameters were collected from predose to up to 24 hours postdose on Day 1 and from predose to up to 72 hours postdose on Day 5 in each treatment period.
Time Frame: Up to 72 hours after study drug administration
Population: Participants with an AUC(0-24hr) measurement
Measure: Mean (Standard Deviation); unit: nmol*hr/L
Groups:
- MK-0941 40mg: Participants receiving MK-0941 40 mg doses three times daily
Arm/Group | MK-0941 5mg | MK-0941 10mg | MK-0941 20mg | MK-0941 40mg
Number analyzed (Participants) | 6 | 7 | 5 | 4
nmol*hr/L
  Day 1 | 754 (165) | 1900 (885) | 3230 (654) | 8700 (2190)
  Day 5 | 883 (157) | 2360 (1260) | 3560 (863) | 9730 (3140)

3. Secondary Outcome: Plasma Pharmacokinetic Parameter: Maximum Concentration (Cmax) of MK-0941
Description: as for outcome 2
Time Frame: Up to 72 hours after study drug administration
Population: Participants with a Cmax measurement
Measure: Mean (Standard Deviation); unit: nmol/L
Arm/Group | MK-0941 5mg | MK-0941 10mg | MK-0941 20mg | MK-0941 40mg
Number analyzed (Participants) | 6 | 7 | 5 | 4
nmol/L
  Day 1 | 105 (21.5) | 255 (116) | 487 (58.3) | 1340 (269)
  Day 5 | 128 (26.2) | 292 (108) | 509 (140) | 1240 (424)

4. Secondary Outcome: Plasma Pharmacokinetic Parameter: Time to Reach Cmax (Tmax) of MK-0941
Description: as for outcome 2
Time Frame: Up to 72 hours after study drug administration
Population: Participants with a Tmax measurement
Measure: Median (Full Range); unit: hr
Arm/Group | MK-0941 5mg | MK-0941 10mg | MK-0941 20mg | MK-0941 40mg
Number analyzed (Participants) | 6 | 7 | 5 | 4
hr
  Day 1 | 3.5 [1.0 to 11.0] | 6.0 [1.0 to 11.0] | 1.0 [1.0 to 6.0] | 1.0 [1.0 to 6.0]
  Day 5 | 1.0 [1.0 to 11.0] | 1.0 [1.0 to 6.0] | 6.0 [6.0 to 11.0] | 6.0 [6.0 to 6.0]

5. Secondary Outcome: Plasma Pharmacokinetic Parameter: Concentration of MK-0941 at 24 Hours (C24hr)
Description: as for outcome 2
Time Frame: Up to 72 hours after study drug administration
Population: Participants with a C24hr measurement
Measure: Mean (Standard Deviation); unit: nmol/L
Arm/Group | MK-0941 5mg | MK-0941 10mg | MK-0941 20mg | MK-0941 40mg
Number analyzed (Participants) | 6 | 7 | 5 | 4
nmol/L
  Day 1 | 8.9 (3.7) | 14.6 (3.7) | 27.9 (12.8) | 66.4 (16.4)
  Day 5 | 9.5 (2.1) | 26.0 (7.4) | 38.5 (12.5) | 112.8 (41.4)

6. Secondary Outcome: Plasma Pharmacokinetic Parameter: Apparent Terminal Elimination Half-life (t1/2) of MK-0941
Description: as for outcome 2
Time Frame: Up to 72 hours after study drug administration
Population: Participants with a t1/2 measurement
Measure: Mean (Standard Deviation); unit: hr
Arm/Group | MK-0941 5mg | MK-0941 10mg | MK-0941 20mg | MK-0941 40mg
Number analyzed (Participants) | 6 | 7 | 5 | 4
hr
  Day 1 | 5.4 (1.5) | 4.4 (1.2) | 4.3 (1.1) | 3.9 (1.1)
  Day 5 | 7.7 (2.0) | 8.3 (4.1) | 9.9 (7.2) | 9.1 (7.3)

7. Primary Outcome: Number of Participants Who Discontinued Study Drug Due to an AE
Description: as for outcome 1
Time Frame: Up to 14 days after last dose of study drug
Population: Safety Population, consisting of all randomized participants who received at least one dose of study drug.
Measure: Number; unit: participants
Arm/Group | Placebo | MK-0941 5mg | MK-0941 10mg | MK-0941 20mg | MK-0941 40mg
Number analyzed (Participants) | 8 | 6 | 6 | 6 | 5
participants | 0 | 0 | 0 | 0 | 0

8. Secondary Outcome: Plasma Pharmacokinetic Parameter: Day 5 to Day 1 Accumulation Ratio for AUC (0-24hr), Cmax, and C24hr
Description: Geometric Mean of the Day 5 to Day 1 Accumulation Ratio
Time Frame: Day 5 and Day 1
Population: All participants with pharmacokinetic measurements on Days 1 and 5
Measure: Geometric Mean (Full Range); unit: Ratio
Arm/Group | MK-0941 5mg | MK-0941 10mg | MK-0941 20mg | MK-0941 40mg
Number analyzed (Participants) | 6 | 7 | 5 | 4
Ratio
  AUC(0-24hr) Day 5/Day 1 Accumulation Ratio | 1.18 [1.09 to 1.38] | 1.28 [1.09 to 1.42] | 1.09 [0.93 to 1.31] | 1.1 [1.04 to 1.22]
  Cmax Day 5/Day 1 Accumulation Ratio | 1.21 [1.05 to 1.42] | 1.18 [0.87 to 1.36] | 1.02 [0.79 to 1.28] | 0.90 [0.72 to 1.08]
  C24hr Day 5/Day 1 Accumulation Ratio | 1.1 [0.61 to 1.96] | 1.77 [1.23 to 2.19] | 1.44 [0.81 to 2.01] | 1.65 [1.07 to 2.61]

ADVERSE EVENTS:
Time Frame: Participants were monitored for occurrence AEs for up to 8 days after last dose of study drug during Period 1 and for up to 14 days after last dose of study drug during Period 2.
Description: This is a crossover-design study; a single participant may be represented in up to two different reporting groups.
Arm/Group | Placebo | MK-0941 5mg | MK-0941 10mg | MK-0941 20mg | MK-0941 40mg
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/6 | 0/6 | 0/6 | 0/5
Other Adverse Events (participants affected / at risk) | 2/8 | 2/6 | 2/6 | 2/6 | 2/5
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=8) | MK-0941 5mg (N=6) | MK-0941 10mg (N=6) | MK-0941 20mg (N=6) | MK-0941 40mg (N=5)
Diabetic retinopathy (Eye disorders) | 1 | 0 | 0 | 0 | 0
Retinopathy (Eye disorders) | 1 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 0 | 2 | 0 | 0 | 0
Wound (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Blood glucose decreased (Investigations) | 0 | 0 | 1 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1 | 1
Headache (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1
Haemorrhage (Vascular disorders) | 0 | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts, or presentations regarding this study 60 days prior to submission for publication/presentation. Any information identified by the SPONSOR as confidential must be deleted prior to submission.